CLINICAL TRIAL: NCT03807206
Title: Resucitation Outcomes in the Netherlands: Flash Mob Research on the Subject of Patient Experiences Regarding Do Not Resuscitate Orders.
Brief Title: Resuscitation Outcomes in the Netherlands Flashmob Questionnaire
Acronym: ROUTINE-F
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: European Society of Anaesthesiology (Other)
Responsible Party: Principal Investigator, Marc Schluep, principal investigator/medical doctor, Erasmus Medical Center
Other Study IDs: ROUTINE-F
Record Dates: First submitted 2019-01-07; First posted 2019-01-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Cardiopulmonary Arrest; DNR-orders
MeSH Terms: conditions — Heart Arrest | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Flashmob 2019: Patients from the following hospitals will receive a questionnaire/structured intereview: Erasmus MC, Franciscus Gasthuis & Vlietland, Ikazia, Haaglanden Medisch Centrum, Albert Schweitzer ziekenhuis, Jeroen Bosch ziekenhuis, Rijnstate ziekenhuis, Amphia ziekenhuis, Tergooi klinieken, Medisch Spectrum Twente, Reinier de Graaf gasthuis. Pending: Maasstad ziekenhuis
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Patient questionnaire
  Other Names: structured interview

SUMMARY:
The aim of this study is to gain insight in patients' experiences regarding do not resuscitate conversations and decisions. A multicentre flash mob investigation will be conducted in which data will be obtained over the course of two weeks using electronic questionnaires that patients will fill out. General demographic data and a brief quality of life assessment (EQ-5D) will be collected. Whether a DNR converstation has taken place will be noted, along with patients' experiences with this conversation. Lastly the patient will be asked about his/her expectations of survival after cardiopulmonary resuscitation.

DETAILED DESCRIPTION:
Rationale: In-hospital cardiac arrest, associated with a survival to discharge of 15.0%, results in a good neurologic discharge in 9.1% - 30.0% of patients. Therefore it is recommended to engage in advanced care planning with patients, to discuss do-not-resuscitate (DNR) directives. In current knowledge, there are no published data about the prevalence of these DNR orders and associated factors in hospitalized patients in the Netherlands. Also, the conversation about DNR are sometimes perceived as awkward or untimely by patients.

Objective: The primary goal is to estimate prevalence DNR order in Dutch hospitals. A secondary goal is to assess what geographical, patient and disease factors are associated with DNR status. Furthermore patient experience in the conversation leading to DNR-orders is of interest.

Study design: A cross-sectional point prevalence study, in 10 participating hospitals of the ROUTiNE project.

Study population: Patients who plan to be admitted for more than 24 hours to the participating hospitals, aged 18 or older, who are responsive and conscious.

Main study parameters/endpoints: The prevalence of DNR orders, expressed as number per 1000 beds.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: There is no risk. Only one ten-minute interview per participant. Therefore the benefit of this study (as described in the objectives) outweigh the potential risks.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the participating hospitals with a planned admission >24 hours at the moment this study takes place.

Exclusion Criteria:

* • Refusal to participate

  * <18 years of age
  * Admitted in outpatient clinic and day treatment centres (e.g. haemodialysis)
  * Admitted <24 hours, as defined by not sleeping overnight in hospital
  * No reliable proxy in the following situations:

    * Unable to answer questions (e.g. unconscious, cognitively impaired, delirious)
    * Language barrier (with no interpreter or family member)
  * The following hospital departments are excluded:

    * Intensive care unit
    * Coronary/acute cardiac care unit
    * Obstetrics
    * Paediatrics
    * Stroke unit
    * Dialysis (outpatient dialysis)
    * Day-care wards/short-stay (i.e. <1 day)
    * Palliative care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The base population consists of all adult patients admitted to all the participating hospitals. These consist of one academic centre and 10 general hospitals. The sampling is based on non-probability as it does not represent the entire population (i.e. inhabitants of the Netherlands), however it is based on probability sampling when the population is solely patients admitted to hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1136 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-02-07 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of DNR-orders | 1 day
  Percentage of DNR-orders in the total cohort as noted in the electronic patient file

SECONDARY OUTCOMES:
DNR-order discussion prevalence | 1 day
  Number of patients who have had a DNR discussion with their physician
DNR-order discussion experience | 1 day
  Patient experience with the DNR-order discussion; was it timely, was the explanation clear?
DNR-order discrepancy | 1 day
  DNR-order reported by the patient, compared to DNR-order from the electronic patient file
Quality of life | 1 day
  EQ-5D (Euroqol): EQ-5D-5L is a standardized, participant-rated instrument for use as a measure of health outcomes. The EQ 5D-5L includes 2 components: the EQ-5D-5L descriptive system and the visual analogue scale (VAS). The EQ-5D-5L descriptive system provides a profile of the participant's health state in 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). For each dimension, the participant is instructed to choose one of 5 levels that best describes their health on that day: "no problem" (1), "slight" (2), "moderate" (3), "severe" (4), or "unable/extreme" (5). The VAS is the participant's rating of their health on a scale of 0 "worst health you can imagine" to 100 "best health you can imagine".

OTHER OUTCOMES:
General demographic data | 1 day
  Demographic profile of inpatients in the Netherlands: age, sex, religion, education, no. of diseases, no. of medications

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jan Stolker, MD PhD, Principal Investigator — Erasmus Medical Center; Monique van Dijk, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (12):
- Netherlands (12):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Rijnstate, Arnhem
  - Amphia, Breda
  - Reinier de Graaf gasthuis, Delft
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Medisch Spectrum Twente, Enschede
  - Tergooi ziekenhuizen, Hilversum
  - Erasmus MC, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - Ikazia, Rotterdam
  - Maasstad, Rotterdam
  - Haaglanden Medisch Centrum, The Hague

IPD SHARING:
Plan to Share IPD: No
Because of the personal nature of data (reg. age, sex, religion, eductional level) we will not make it available.